CLINICAL TRIAL: NCT06614556
Title: Quantifying the Trainability of Peripheral Nerve Function in Young and Older Adults.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oklahoma State University (Other)
Collaborators: American College of Sports Medicine - Central States Chapter (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: IRB-22-270
Record Dates: First submitted 2024-09-12; First posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Nerve Degeneration; Healthy Aging
MeSH Terms: conditions — Nerve Degeneration | interventions — Resistance Training; Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Young Training Group (Experimental): Ages 18-35. Performed 4 weeks of an at-home, hand grip resistance training intervention.
  Interventions: Other: Resistance Training
- Young Control Group (No Intervention): Ages 18-35. Did not perform the training intervention
- Older Training Group (Experimental): Ages 60+. Performed 4 weeks of an at-home, hand grip resistance training intervention.
  Interventions: Other: Resistance Training
- Older Control Group (No Intervention): Ages 60+. Did not perform the training intervention

INTERVENTIONS:
Other: Resistance Training — Participants in the training groups performed bilateral hand grip resistance training three times per week for four weeks using a specialized hand-grip kit provided to them. Participants were provided with pictures and instructions for each exercise upon completion of the initial testing (PRE) session. They were asked to perform 12 training sessions (approximately 30-45 mins) over the 4 weeks according to their schedule. Each participant was asked to keep a training log to assist with accountability. Those assigned to the control groups were asked to maintain their normal daily activities throughout the four weeks.
  Other Names: Strength Training; Exercise
  Arms: Older Training Group; Young Training Group

SUMMARY:
The purpose of this project is to identify the effects of hand grip resistance training on nerve speed of the hand muscles and to quantify whether age plays a role in those effects. Two groups (young and older adults) underwent a 4-week resistance training intervention with nerve conduction velocity measured before and after. There were also two control groups (young and older adults) who performed the testing 4 weeks apart, but did not engage in the intervention.

DETAILED DESCRIPTION:
Studies have shown that nerve speed slows with advancing age. As a result, slower nerves may result in slower movement speed and can alter response time. The investigators propose that a resistance training intervention may elicit positive adaptations to the nerves. The purpose of this project is to identify the effects of hand grip resistance training on nerve speed of the hand muscles and to quantify whether age plays a role in those effects. Two groups (young and older adults) underwent a 4-week, at-home, resistance training intervention with nerve conduction velocity (m/s) measured before and after. There were also two control groups (young and older adults) who performed the testing 4 weeks apart, but did not engage in the intervention. Other outcome measures included nerve size, via ultrasound, maximal handgrip strength, and hand dexterity.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy adults 18 - 100 years old.

Exclusion Criteria:

* If you have been notified by a physician to refrain from exercise due to cardiovascular issues.
* Known orthopedic or neuromuscular limitations or illness of the upper extremities.
* Known neuromuscular disorders.
* Individuals that are experiencing a fever (> 100.4° F) or have identified as symptomatic on the COVID-19 screening questionnaire may not participate at this time.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2022-09-20 (Actual); Primary Completion 2023-07-18 (Actual); Study Completion 2023-07-18 (Actual)

PRIMARY OUTCOMES:
Motor nerve conduction velocity (m/s) | Before and after 4 weeks of training (or just 4 weeks, for controls)
  Conduction velocity of the median nerve, via nerve stimulation, as measured through EMG at the Flexor Digitorum Superficialis muscle

SECONDARY OUTCOMES:
Nerve cross-sectional area (mm^2) | Before and after 4 weeks of training (or just 4 weeks, for controls)
  The area within the visible borders of the nerve, as seen and measured via ultrasound
Maximal strength (kg) | Before and after 4 weeks of training (or just 4 weeks, for controls)
  Maximal handgrip strength using a handgrip dynamometer
Hand motor dexterity (seconds) | Before and after 4 weeks of training (or just 4 weeks, for controls)
  A timed Minnesota manual dexterity task

CONTACTS AND LOCATIONS:
Overall Officials: Jason M DeFreitas, PhD, Principal Investigator — Oklahoma State University
Locations (1):
- Applied Neuromuscular Physiology Laboratory, Stillwater, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-09-17): https://cdn.clinicaltrials.gov/large-docs/56/NCT06614556/Prot_SAP_000.pdf
  • Informed Consent Form (2024-09-09): https://cdn.clinicaltrials.gov/large-docs/56/NCT06614556/ICF_001.pdf